CLINICAL TRIAL: NCT03521973
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess Safety, Tolerability and Protective Efficacy of PfSPZ Vaccine in 1-12 Year-old Gabonese Children Naturally Exposed to Malaria Parasites
Brief Title: Safety, Tolerability and Protective Efficacy of PfSPZ Vaccine in Gabonese Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Centre de Recherches Médicales de Lambaréné (CERMEL), German Center for Infection Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LaSPZV1
Record Dates: First submitted 2018-04-26; First posted 2018-05-11 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1- PfSPZ-Vaccine (Experimental): Children aged 7-12 years (inclusive) of age will be enrolled in this group.
  N=44 will receive PfSPZ Vaccine; three doses of 9x10^6 PfSPZ of PfSPZ Vaccine administered by direct venous inoculation (DVI) given at 0, 7 and 28 day intervals.
  Interventions: Biological: PfSPZ Vaccine
- Group 2 (Placebo Comparator): Children aged 7-12 years (inclusive) of age will be enrolled in this group.
  N=22 will receive normal saline; three doses of NS administered by DVI given at 0, 7 and 28 day intervals.
  Interventions: Other: Normal Saline
- Group 3 (Experimental): Children aged 3-6 years (inclusive) of age will be enrolled in this group.
  N=44 will receive PfSPZ Vaccine; three doses of 9x10^6 PfSPZ of PfSPZ Vaccine administered by direct venous inoculation (DVI) given at 0, 7 and 28 day intervals; given 2 weeks after the first immunization of Group 1.
  Interventions: Biological: PfSPZ Vaccine
- Group 4 (Placebo Comparator): Children aged 3-6 years (inclusive) of age will be enrolled in this group.
  N=22 will receive normal saline; three doses of NS administered by DVI given at 0, 7 and 28 day intervals; given 2 weeks after the first dose of NS of Group 2.
  Interventions: Other: Normal Saline
- Group 5 (Experimental): Children aged 1-2 years (inclusive) of age will be enrolled in this group.
  N=44 will receive PfSPZ Vaccine; three doses of 9x10^6 PfSPZ of PfSPZ Vaccine administered by direct venous inoculation (DVI) given at 0, 7 and 28 day intervals; given 2 weeks after the first immunization of Group 3.
  Interventions: Biological: PfSPZ Vaccine
- Group 6 (Placebo Comparator): Children aged 1-2 years (inclusive) of age will be enrolled in this group.
  N=22 will receive normal saline; three doses of NS administered by DVI given at 0, 7 and 28 day intervals; given 2 weeks after the first dose of NS of Group 4.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Radiation-attenuated, aseptic, purified, cryopreserved Plasmodium falciparum sporozoites (PfSPZ Vaccine)
  Arms: Group 1- PfSPZ-Vaccine; Group 3; Group 5
Other: Normal Saline — 0.9% Sodium chloride
  Other Names: NS
  Arms: Group 2; Group 4; Group 6

SUMMARY:
This study is a single site, randomized, double-blind, placebo-controlled trial. The trial will assess the safety, tolerability, immunogenicity and vaccine efficacy (VE) of PfSPZ Vaccine in Gabonese children that are naturally exposed to malaria parasites. Healthy children aged 1- 12 years living in the surrounding areas of Lambaréné and/or Fougamou Province in Gabon will be eligible for participation.

DETAILED DESCRIPTION:
The trial will be performed in 200 healthy Gabonese children, recruited across three age-strata: 7-12, 3-6 and 1-2 years (12-35 months). Within each age-stratum, volunteers will be randomized in a 2:1 ratio to receive three doses via direct venous inoculation (DVI) of either PfSPZ Vaccine (0.9x10^6) or normal saline (NS) on days 0, 7 and 28 respectively; a minimum of 40 and a maximum of 100 volunteers are included in each of these age-strata.

In total, approximately 133 children will receive PfSPZ Vaccine and approximately 67 children will receive placebo. Randomization will be stratified by age-stratum, using permuted blocks of randomized size (3, 6, or 9). The start of inclusion into each age-stratum will be staggered, such that immunization of the first 3-6-year-olds will not commence until two weeks after start of immunization in the first 7-12-year-olds, and immunizations in the first 1-2-year-olds will not commence until two weeks after start of immunization in the first 3-6-year-olds. All volunteers will receive presumptive treatment with artemether-lumefantrine two weeks prior to final immunization (day 14). All volunteers will receive presumptive treatment with age-standardized 3-day course of oral artemether-lumefantrine (AL) ~two weeks prior to first immunization and again two weeks prior to final immunization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 1 to 12 years
* Provision of written informed consent of a legal representative of age 18 or above and provision of informed assent by participants in concordance with Gabonese national guidelines.
* Able and willing to comply with all study requirements
* Residence in the area throughout the study period
* Household member reachable by mobile phone during the immunization phase

Exclusion Criteria:

* Receipt of an investigational product in the 30 days preceding enrollment
* Prior receipt of a malaria vaccine
* Immunization with more than 3 other vaccines or at least on elive vaccine within the past four weeks
* Use of immunoglobulins or blood products within 3 months prior to immunization with the investigational product
* Known or suspected HIV infection or any other immunosuppressive state
* Positive for hepatitis B surface antigen (HBs-antigen)
* Seropositive for hepatitis C virus (antibodies to HCV)
* A hemoglobin concentration <9 g/dl (applies at enrollment only)
* History of non-febrile or atypical febrile seizures
* Pregnancy or lactation
* Any other significant disease, disorder or finding which, in the opinion of the investigator, may significantly increase the risk to the child because of participation in the study or impair interpretation of the study data

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers who become parasitemic will be recorded, detected by Thick Blood Smear (TBS) microscopy | From 2 weeks to 6 months after the third PfSPZ Vaccine immunization
  Time to event and proportional analysis of episodes of P. falciparum parasitemia, detected actively or passively by TBS microscopy. Vaccine efficacy will be measured in the mITT population.
Proportion of volunteers who become parasitemic with temperature ≥37.5°C or history of fever | From 2 weeks to 6 months after the third PfSPZ Vaccine immunization
  Time to event and proportional analysis of episodes of P. falciparum parasitemia with temperature ≥37.5°C or history of fever within the last 24 hours (P. falciparum malaria with clinical manifestations). Vaccine efficacy against P. falciparum malaria with clinical manifestations will be measured in the mITT population using hierarchical testing; the secondary will only be tested when the primary endpoint shows a significant difference.
The occurrence and frequency of adverse events (AEs) | From the time of each PfSPZ Vaccine immunization until 7 days after each dose
  The occurrence and frequency of Grade 3 solicited adverse AEs (related or unrelated) after vaccination
The occurrence and frequency of AEs | From the time of first PfSPZ Vaccine immunization until 28 days after the last dose
  The occurrence and frequency of Grade 3 unsolicited adverse AEs (related or unrelated) after vaccination
The occurrence and frequency of serious adverse events (SAEs) | Around 27 months (from day of first immunization through study completion)
  The occurrence and frequency of SAEs (related or unrelated) after vaccination

SECONDARY OUTCOMES:
The occurrence of all related solicited AE | From the time of each PfSPZ Vaccine immunization until 7 days after each dose
  The occurrence of all related solicited AE after vaccination
The occurrence of all related unsolicited AEs | From the time of first PfSPZ Vaccine immunization until 28 days after the last dose
  The occurrence of all related unsolicited AE after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Selidji Agnandji, MD, Principal Investigator — Centre de Recherches Médicales de Lambaréné (CERMEL)
Locations (1):
- Centre de Recherches Médicales de Lambaréné (CERMEL), Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Derived] Agnandji ST, Bok J, Alabi A, Kabwende AL, Mbouna A, Bie J, Moukiti E, Lalremruata A, Esen M, Kreidenweiss A, Kc N, Sim BKL, Richie TL, Preston Church LW, McCall MBB, Hoffman SL, Kremsner PG, Mordmuller B. Safety, tolerability, and protective efficacy of a radiation-attenuated, whole sporozoite malaria vaccine in children in Gabon: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2026 Jan;26(1):79-90. doi: 10.1016/S1473-3099(25)00434-7. Epub 2025 Sep 16. PMID 40972633